CLINICAL TRIAL: NCT06342999
Title: Evaluation of Outcomes of Fetal Aortic Valvuloplasty for Evolving Hypoplastic Left Heart Syndrome
Brief Title: Fetal Aortic Valvuloplasty for Evolving Hypoplastic Left Heart Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mauro H. Schenone (Other)
Responsible Party: Sponsor-Investigator, Mauro H. Schenone, Regulatory Sponsor and Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-012399
Record Dates: First submitted 2024-03-27; First posted 2024-04-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hypoplastic Left Heart Syndrome
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group: Fetal Aortic Valvuloplasty (Experimental): Women diagnosed with HLHS will undergo fetal aortic valvuloplasty between 21 and 29 weeks gestation.
  Interventions: Procedure: Fetal Aortic Valvuloplasty Procedure; Device: Emerge Monorail and Over-The-Wire PTCA Dilatation Catheter; Device: Trek RX and Mini Trek RX Coronary Dilatation Catheter
- Control Group: Expectant Management (No Intervention): Women diagnosed with HLHS will undergo expectant management with postnatal surgery.

INTERVENTIONS:
Procedure: Fetal Aortic Valvuloplasty Procedure — Treatment given during pregnancy in which a balloon is used to increase the size of the baby's aortic valve in vitro.
  Arms: Intervention Group: Fetal Aortic Valvuloplasty
Device: Emerge Monorail and Over-The-Wire PTCA Dilatation Catheter — Balloon Catheter
  Arms: Intervention Group: Fetal Aortic Valvuloplasty
Device: Trek RX and Mini Trek RX Coronary Dilatation Catheter — Coronary Dilation Catheter
  Arms: Intervention Group: Fetal Aortic Valvuloplasty

SUMMARY:
The purpose of this research is to investigate the best way to manage evolving hypoplastic left heart syndrome (HLHS).

DETAILED DESCRIPTION:
The condition occurs when part of the heart doesn't develop properly so the heart is not able to pump blood around the body effectively. Babies born with this condition require surgery and are often left with a lifelong heart disability. A number of babies with this condition will die during pregnancy or within the first year of life (approximately 10-40%). We are investigating a treatment given during pregnancy in which a balloon is used to increase the size of the baby's aortic valve. The aortic valve function is to allow easy flow from the heart to the body and prevent blood from returning to the heart (regurgitation). This is called fetal aortic valvuloplasty. A number of studies have shown promising results, including a higher of the baby surviving with both sides of the heart functioning (as opposed to only the right side), this may also lead to longer survival with a better quality of life. However, we do not have enough information to say this is always the best way to manage the condition. Currently, parents of babies with this condition, who meet certain eligibility criteria, are offered fetal aortic valvuloplasty during pregnancy. The alternative option is not to intervene during pregnancy but instead monitor the baby with regular ultrasounds. We call this conservative management.

ELIGIBILITY:
Inclusion Criteria

* Pregnant women 18-45 years of age.
* Gestational age between 21 0/7 and 29 6/7 weeks of gestation
* The mother must be healthy enough to undergo surgery.
* The individual being enrolled must be able to provide informed consent.
* Dominant cardiac defect is valvar
* Evolving hypoplastic left heart syndrome defined as depressed left ventricle systolic and at least one of the following:

  * Retrograde flow in the transverse aortic arch
  * Two of the following: (1) left to right flow across the atrial septum (bulging of the septum left to right in cases of intact atrial septum); (2) monophasic mitral valve inflow; (3) bidirectional flow in the pulmonary veins.
* Potential for a technically successful and postnatal biventricular outcome defined as left ventricle long axis Z-score equal or greater than -2 PLUS at least 4 of the following 5 criteria:

  * Left ventricle long axis Z-score more than zero
  * Left ventricle short axis Z-score more than zero
  * Aortic annulus Z-score more than -3.5
  * Mitral valve annulus Z-score more than -2
  * Left ventricle generating a maximal instantaneous gradient (MIG) equal or greater than 20 mmHg (or by mitral regurgitation jet greater than or equal to 20 mmHg).

Exclusion Criteria

* Patient is less than 18 years of age or more than 45 years of age.
* Contraindication to anesthesia or surgery
* Preterm labor or cervical length <20 mm at enrollement or uterine anomaly strongly predisposing to preterm delivery.
* Other fetal anomalies that significantly impact fetal/neonatal survival (e.g., congenital diaphragmatic hernia, bilateral renal agenesis, etc.)
* Fetal aneuploidy and pathogenic findings on Karyotype or Microarray that impact significantly the fetal/neonatal survival.
* Cases with all the following criteria:

  * Left ventricle pressure ≤ 47 mmHg
  * MV dimension Z-score < 0.1
  * MV inflow time Z-score < -2

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2036-07 (Estimated); Study Completion 2036-07 (Estimated)

PRIMARY OUTCOMES:
Number of cases in which the procedure was successful | Baseline
  Procedure success defined as the aortic valve was crossed and the balloon inflated with clear evidence of improvement of blood flow through the aortic valve and or new aortic valve regurgitation
Number of cases in which a biventricular repair was achieved | Baseline
Number cases with pulmonary hypertension | Baseline

SECONDARY OUTCOMES:
Number of cases delivered prematurely | Baseline
Number of cases with perinatal death | Baseline
Number of maternal complications | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Schenone, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials